CLINICAL TRIAL: NCT05123534
Title: A Phase 2 Dose-escalation Study Examining the Safety, Pharmacokinetics, and Preliminary Efficacy of Ascending Drug and Energy Dose Combinations for Sonodynamic Therapy Using SONALA-001 in Combination with Exablate 4000 Type 2.0 MR-Guided Focused Ultrasound in Subjects with Diffuse Intrinsic Pontine Glioma (DIPG) and Diffuse Midline Glioma (DMG)
Brief Title: A Phase 2 Study of Sonodynamic Therapy Using SONALA-001 and Exablate 4000 Type 2.0 in Patients with DIPG
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: The study is suspended due to lack of funding but not due to safety concerns.
Sponsor: SonALAsense, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SDT-201; FD-R-7538 (Other Grant/Funding Number: FDA OOPD); R44CA261516 (NIH)
Record Dates: First submitted 2021-10-11; First posted 2021-11-17 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Diffuse Intrinsic Pontine Glioma; Diffuse Midline Glioma
Keywords: DIPG; Sonodynamic Therapy; Exablate 4000 Type 2.0; MR-guided Focused Ultrasound; SONALA-001; SDT; MRgFUS; Aminolevulinic acid HCI; ALA HCI; ALA; DMG
MeSH Terms: conditions — Diffuse Intrinsic Pontine Glioma

STUDY DESIGN:
Intervention Model Description: Drug/energy dose escalation to identify the RP2D as guided by BOIN for the combination of SONALA-001 and Exablate 4000 Type 2.0 MRgFUS.
  The primary focus of the proposed study is safety, tolerability and determination of the MTD and RP2D; therefore, statistical modeling and inferential statistics are not planned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (5):
- Cohort 1 (Experimental): 5 mg/kg IV SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy Level 1
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Cohort 2 (Experimental): 5 mg/kg IV SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy Level 2
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Cohort 3 (Experimental): 10 mg/kg IV SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy Level 3
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Cohort 4 - DIPG Cohort at RP2D (Experimental): The RP2D of SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)
- Cohort 5 - DMG Cohort at RP2D (Experimental): The RP2D of SONALA-001 (ALA) and MR-guided Focused Ultrasound (MRgFUS) Energy
  Interventions: Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS)

INTERVENTIONS:
Combination Product: SONALA-001 (ALA) and MR-Guided Focused Ultrasound device (MRgFUS) — SONALA-001(ALA) given 6-12 hours prior to receiving the MRgFUS.
  Other Names: Exablate Type 2.0

SUMMARY:
The primary objectives of this trial are to evaluate the safety and tolerability of sonodynamic therapy (SDT) using SONALA-001 and Exablate Type 2.0 device and to determine the maximum tolerated dose (MTD) or recommended phase 2 dose (RP2D) of MR-Guided Focused Ultrasound (MRgFUS) energy in combination with SONALA-001 in subjects with diffuse intrinsic pontine glioma

Funding Source - FDA OOPD

ELIGIBILITY:
Inclusion Criteria:

DIPG Subjects:

1. Newly diagnosed, radiographically typical DIPG, defined as a tumor with a pontine epicenter and diffuse involvement of more than ⅔ of the pons and without evidence of dissemination, are eligible with or without histologic confirmation.

   * The diagnosis imaging scan must be reviewed by the study site's neuroradiologist and the principal investigator. The diagnosis imaging scan must subsequently be sent to the study central imaging vendor.
   * Subjects who present with DIPG and dissemination at diagnosis, but after completion of radiotherapy have no dissemination on neuroimaging at screening, are considered eligible.
   * Subjects with pontine lesions that do not meet radiographic criteria will be eligible if there is histologic confirmation of DIPG.
   * Subjects may be asked to agree to provide access to previously obtained biopsy results.
   * If tumor status is unknown or archival tumor tissue is not available, subjects may be asked to agree to submit a post-mortem biopsy specimen to enable molecular profiling of tumor.
2. Prior treatment consisting of a minimum of 54 Gy standard focal radiotherapy administered over 42-49 days.
3. Must be ≥ 4 weeks and ≤ 24 weeks post radiotherapy and must have recovered from acute effects to CTCAE (version 5) Grade 1 or baseline prior to Day 1.
4. Must have stable to improved imaging by RAPNO (subjects ≤ 21 years of age) and mRANO (subjects > 21 years of age) criteria comparing the scan obtained post radiotherapy to the scan obtained during the screening period. The comparison of diagnosis imaging scan and screening imaging scan must be reviewed by the study site's neuroradiologist and the principal investigator. If subjects present within 3 months after completion of radiotherapy and the comparison of the diagnosis scan to the screening scan is consistent with RAPNO/mRANO progression but pseudoprogression is a consideration, then the subject can be re-screened if the subject falls out of the screening window.
5. Subjects who are on steroids must be on a stable to decreasing dose of steroids (maximum dexamethasone of 1 mg/m2/day) prior to Day 1.
6. Minimum of 5 years of age. Subjects younger than 5 years old may be eligible after discussion with the Sponsor Medical Monitor/designee.
7. A minimum head circumference of 52 cm as measured by physical exam. Subjects with a minimum head circumference smaller than 52 cm may be eligible after discussion with the Sponsor Medical Monitor/designee.
8. Females of childbearing potential (FOCP) must have a negative serum or urine pregnancy test at screening. Subjects of childbearing or child fathering potential must be willing to use highly effective birth control during the entire study. Acceptable forms of birth control include hormonal contraceptives (oral, injectable, transdermal, or intravaginal) or intrauterine device (IUD) for at least one week prior to ALA SDT, condom and spermicidal or diaphragm and spermicidal. Other acceptable forms of birth control include a) abstinence for subjects who are not sexually active; or b) if the subject is in a monogamous relationship with a partner who is sterile (e.g., vasectomy performed at least 6 months prior to subject's ALA SDT treatment). Subjects who become sexually active or begin to have relations with a partner who is not sterile during the trial must agree to use an effective form of birth control for the duration of the study. FOCP taking hormonal therapy must be on treatment for at least 12 weeks prior to study entry and must not change their dosing regimen during the study.
9. Ability to provide written, signed, and dated (personally or via a legally authorized representative) informed consent/and assent at screening as applicable to participate in the study.
10. Karnofsky Performance Scale (KPS for > 16 years of age) or Lansky Performance Score (LPS for ≤ 16 years of age) assessed within 14 days of Day 1 must be ≥ 50%. Subjects who are unable to walk because of neurologic deficits, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
11. Subjects must have adequate organ and marrow function as defined below:

    * Absolute neutrophil count ≥ 1,000/mm3, without the use of myeloid growth factors (e.g. GCSF) within 7 days prior to Day 1.
    * Platelets ≥ 100,000/mm3 (unsupported, defined as no platelet transfusion within 7 days prior to Day 1).
    * Hemoglobin ≥ 8 g/dl maintained without the need for erythropoietin stimulating agents (may have received last transfusion within 7 days prior to Day 1).
    * Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN); in subjects with Gilbert syndrome, total bilirubin >1.5 ULN as long as direct bilirubin is normal.
    * Alanine aminotransferase (ALT) < 3 x institutional ULN.
    * Aspartate aminotransferase (AST) < 3 x institutional ULN.
    * Albumin ≥ 3 g/dl.
    * Potassium ≥ lower limit of normal (LLN).
    * Serum total calcium (correct for serum albumin) or ionized calcium ≥ LLN.
    * Renal function as defined below:

      * Age 5-17 years: GFR ≥ 70 mL/min/1.73m2 as estimated by Schwartz formula (Schwartz, 2009). If eGFR is abnormal for age based on Schwartz formula, accurate measurement should be obtained by 24-hour creatinine clearance (CrCl).
      * Age ≥ 18 years: CrCl ≥ 60 mL/min/1.73m2 as estimated by the Cockcroft-Gault (C-G) equation. If estimated CrCl is abnormal, accurate measurement should be obtained by 24 hour CrCl.
12. Cardiac function as defined below:

    * Left ventricular ejection fraction ≥ 50% by gated radionuclide study OR shortening fraction of ≥ 27% by echocardiogram.
    * Presence of no ventricular arrhythmias except for benign premature ventricular contractions.
    * QTcF (Fridericia) interval < 450 ms.
13. All colony-forming growth factor(s) (i.e., filgrastim, sargramostim, or erythropoietin) must have been discontinued for at least 7 days prior to Day 1 or 14 days if PEG formulations were received.
14. An understanding, ability, and willingness to fully comply with study procedures and restrictions.
15. Subjects with Ommaya Reservoirs, VP shunts (nonmetallic) or similar will have a technical evaluation of the screening non-contrast CT scan of the head conducted by an Insightec trained technical Research and Development (R&D) specialist which will be provided to SonALAsense. This information will be included in the eligibility review by SonALAsense and designee. During mapping of the target area, if the machine determines that it cannot treat within the safety limits of the system (i.e., skull area, number of elements, etc.), the device will signal that it cannot initiate a sonication at that target and the investigator will determine whether to proceed with the treatment.

DMG Subjects:

1. Age ≥ 5 years old. Subjects younger than 5 years old may be eligible after discussion with the Sponsor Medical Monitor/designee.
2. Radiological diagnosis of Diffuse Midline Glioma (DMG) with tumor involving the pons (intrinsic, pontine based infiltrative lesion; hypointense on T1 weighted images (T1WIs) and hyperintense in T2 sequences, with mass effect on the adjacent structures and occupying at least 50% of the pons), thalami, cerebellum, and/or molecular confirmation of H3K27M mutation of pontine, thalamic, cerebellar glioma.
3. Subjects may be asked to agree to provide access to previously obtained biopsy results.
4. Prior treatment consisting of institutional standard of radiotherapy (including the combination with chemotherapy, by institutional standard) that was completed ≥ 4 weeks and ≤ 24 weeks prior to Day 1, and must have recovered from acute effects to CTCAE (version 5) Grade 1 or baseline prior to Day 1.
5. Subjects who recur/progressed after tumor resection are not excluded.
6. Must have stable to improved imaging by RAPNO/mRANO criteria comparing the scan obtained post radiotherapy to the scan obtained during the screening period. The comparison of diagnosis imaging scan and screening imaging scan must be reviewed by the study site's neuroradiologist and the principal investigator. If subjects present within 3 months after completion of radiotherapy and the comparison of the diagnosis scan to the screening scan is consistent with RAPNO/mRANO progression but pseudoprogression is a consideration, then the subject can be re-screened if the subject falls out of the screening window.
7. Subjects who are on steroids must be on a stable to decreasing dose of steroids prior to Day 1, with a maximum dexamethasone of 1 mg/m²/day, pediatric or adult population or by institutional standard.
8. Performance status assessed within 14 days of Day 1: Karnofsky (age ≥ 16 years) or Lansky (age < 16) score ≥ 50% allowing for stable neurological deficit due to DMG.
9. Subjects must have fully recovered from the acute toxic effects of all prior anti-cancer therapy prior to Day 1 and must meet the following minimum duration from prior anti- cancer directed therapy prior to enrollment.

   • Stem cell infusions: at least 42 days must have elapsed after completion of an autologous stem cell infusion, and at least 84 days must have elapsed after completion of an allogeneic stem cell infusion.
10. Cellular therapy: at least 42 days must have elapsed since the completion of any type of cellular therapy.
11. Subjects must have adequate organ and marrow function as defined below:

    * Absolute neutrophil count ≥ 1,000/mm³, without the use of myeloid growth factors (e.g., GCSF) within 7 days prior to Day 1.
    * Platelets ≥ 100,000/mm³ (unsupported, defined as no platelet transfusion within 7 days prior to Day 1).
    * Hemoglobin ≥ 8 g/dl maintained without the need for erythropoietin stimulating agents (may have received last transfusion within 7 days prior to Day 1).
    * Total bilirubin ≤ 1.5 times institutional upper limit of normal (ULN); in subjects with Gilbert syndrome, total bilirubin >1.5 ULN as long as direct bilirubin is normal.
    * ALT < 3 x institutional ULN.
    * AST < 3 x institutional ULN.
    * Albumin ≥ 3 g/dl.
    * Potassium ≥ lower limit of normal (LLN).
    * Serum total calcium (correct for serum albumin) or ionized calcium ≥ LLN.
    * Renal Function as defined below:

      * Age 5-17 years: GFR ≥ 70 mL/min/1.73 m² as estimated by Schwartz formula (Schwartz, Munoz et al. 2009). If eGFR is abnormal for age based on Schwartz formula, accurate measurement should be obtained by 24-hour creatinine clearance (CrCl).
      * Age ≥ 18 years: CrCl ≥ 60 mL/min/1.73 m² as estimated by the Cockcroft- Gault (C-G) equation. If estimated CrCl is abnormal, accurate measurement should be obtained by 24-hour CrCl.
12. Cardiac Function as defined below:

    * Left ventricular ejection fraction ≥ 50% by gated radionuclide study OR shortening fraction of ≥ 27% by echocardiogram.
    * Presence of no ventricular arrhythmias except for benign premature ventricular contractions.
    * QTcF (Fridericia) interval < 450 ms.
13. All colony-forming growth factor(s) (i.e., filgrastim, sargramostim or erythropoietin) must have been discontinued for at least 7 days prior to Day 1 or 14 days if PEG formulations were received.
14. Subjects with Ommaya Reservoirs, VP shunts (nonmetallic) or similar will have a technical evaluation of the screening non-contrast CT scan of the head conducted by an Insightec trained technical R&D specialist which will be provided to SonALAsense. This information will be included in the eligibility review by SonALAsense and designee. During mapping of the target area, if the machine determines that it cannot treat within the safety limits of the system (i.e., skull area, number of elements, etc.), the device will signal that it cannot initiate a sonication at that target and the investigator will determine whether to proceed with the treatment.
15. Ability to provide written, signed, and dated (personally or via a legally authorized representative) informed consent/and assent at screening as applicable to participate in the study.

Exclusion Criteria:

DIPG Subjects:

1. Evidence of progressive disease by radiologic criteria (RAPNO for subjects ≤ 21 years of age or mRANO for subjects > 21 years of age).
2. Increasing steroid dose prior to Day 1.
3. Diagnosis of porphyria.
4. Hypersensitivity against porphyrins.
5. Current malignancies or relevant history of other malignancy, physical, or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
6. Known history of human immunodeficiency virus (HIV), hepatitis B or C infection, or any active systemic infection.
7. Use of potentially phototoxic substances (e.g., St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, tetracyclines, sulfonamides, quinolones, hypericin extracts, topical preparations containing ALA) within 24 hours before and after SONALA-001 infusion.
8. Prior or concurrent therapy with any other anticancer (including radiotherapy, with the exception of radiotherapy administered per inclusion criteria #2 and #3) or investigational drug or other investigational intervention. NOTE: The use of bevacizumab or similar agent to control radiation therapy-induced edema is allowed for up to a maximum of 5 doses. The last dose must have been administered no later than 14 days prior to Day 1. See Section 6 (Prior and Concomitant Treatment) for a list of prohibited and restricted medications.
9. Use of fish oil supplements within 24 hours of Day 1 is allowed if the subject's clotting parameters fall within normal limits.
10. Use of blood thinning agents within 7 days prior to Day 1. Subjects whose medical condition does not permit discontinuation of this therapy are excluded.
11. Significant acute deterioration in neurologic status within 7 days prior to Day 1, in the opinion of the investigator.
12. Inability to undergo MRI (e.g., presence of a pacemaker).
13. Pregnancy or breastfeeding.
14. Inability to return to study site for required study treatment and follow-up visits (i.e., due to residing or traveling outside of the United States). This includes inability to have local follow-up visits as allowed and outlined per protocol.
15. Metal devices including but not limited to implanted devices in the brain or skull (e.g., shunts, catheters, drains, implants, clips, or other metallic implanted objects) are not allowed. NOTE: Ommaya Reservoirs, VP shunts (non-metallic) or similar are allowed.
16. A known or underlying medical condition that, in the opinion of the investigator or Sponsor, could make the administration of investigational drug/study treatment hazardous to the subject, or could adversely affect the ability of the subject to comply with or tolerate the study.

DMG Subjects:

1. Increasing steroid dose prior to Day 1.
2. Diagnosis of porphyria.
3. Hypersensitivity against porphyrins.
4. Current malignancies or relevant history of other malignancy, physical, or psychiatric illness, any medical disorder that may require treatment or make the subject unlikely to fully complete the study, or any condition that presents undue risk from the investigational product or procedures.
5. Known history of human immunodeficiency virus (HIV), hepatitis B or C infection, or any active systemic infection.
6. Use of potentially phototoxic substances (e.g., St. John's wort, griseofulvin, thiazide diuretics, sulfonylureas, phenothiazines, tetracyclines, sulfonamides, quinolones, hypericin extracts, topical preparations containing ALA) within 24 hours before and after SONALA-001 infusion.
7. Prior or concurrent therapy with any other anticancer therapy with the exception of radio-chemotherapy and stem cell and cellular therapy administered for DMG as described in inclusion criteria NOTE: The use of bevacizumab or similar agent to control radiation therapy-induced edema is allowed for up to a maximum of 5 doses. The last dose must have been administered no later than 14 days prior to Day 1.
8. Use of fish oil supplements within 24 hours of Day 1 is allowed if the subject's clotting parameters fall within normal limits.
9. Use of blood thinning agents within 7 days prior to Day 1. Subjects whose medical condition does not permit discontinuation of this therapy are excluded.
10. Significant acute deterioration in neurologic status within 7 days prior to Day 1, in the opinion of the investigator.
11. Pregnancy or breastfeeding.
12. Inability to return to study site for required study treatment and follow-up visits (i.e., due to residing or traveling outside of the United States). This includes the inability to have local follow-up visits as allowed and outlined per protocol.
13. Inability to undergo MRI (e.g., presence of a pacemaker) or presence of metal devices that are not MRI compatible, including but not limited to implanted devices in the brain or skull (e.g., shunts, catheters, drains, implants, clips, or other metallic implanted objects) are not allowed. NOTE: Ommaya Reservoirs, VP shunts (non-metallic) or similar are allowed.
14. A known or underlying medical condition that, in the opinion of the investigator or Sponsor, could make the administration of investigational drug/ study treatment hazardous to the subject, or could adversely affect the ability of the subject to comply with or tolerate the study.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of SDT in DIPG subjects to generate data that will aid in the design of a larger Phase 2b trial. | Day 1 (SDT Study Treatment Day) to 12 months post-treatment
  Safety and tolerability as assessed by the frequency and severity of dose-limiting toxicities (DLTs), AEs, laboratory and ECG tests, vital signs, weight, physical and neurological exams.
To determine the Maximum Tolerated Dose (MTD) or Recommended Phase 2 Dose (RP2D) of MR-Guided Focused Ultrasound (MRgFUS) energy in combination with SONALA-001 (SDT) in subjects with DIPG. | Up to 3 weeks post-treatment
  MTD and RP2D (determined in consultation with the Safety Review Committee [SRC]): The Bayesian Optimal Interval (BOIN) (SONALA-001 and MRgFUS) method will be employed to derive an MTD for the combination drug and device and estimate RP2D. "R Package for Designing Single-Agent and Drug-Combination Dose-Finding Trials Using Bayesian Optimal Interval Designs" will be implemented.

SECONDARY OUTCOMES:
Preliminary efficacy, including objective response rate (ORR); Response Assessment in Pediatric Neuro-Oncology (RAPNO); Modified Response Assessment in Neuro-Oncology (mRANO). | Day 1 to 12 months
  Objective Response Rate ([ORR], RAPNO or mRANO Criteria): An estimate of RAPNO-ORR or mRANO-ORR, dependent on the age of the subject, will be derived as the percentage of subjects achieving a complete or partial response (CR, PR) relative to the total sample size in the full analysis set.
Progression-free survival (PFS) | Day 1 to 12 months
  PFS is defined as the time from enrollment to the first progressive disease or all-cause mortality.
Duration of response (DOR) | Day 1 to 12 months
  The time-to-event under consideration in the analysis of DOR will be time from onset of (RAPNO) response to the time of first progression of disease.
Overall survival (OS) | Day 1 to 24 months
  OS is defined as the time from enrollment to all-cause mortality.
To evaluate the pharmacokinetics (PK) of ALA and Protoporphyrin IX (PpIX) following intravenous (IV) dosing with SONALA-001. | Day 1 to 24 hours post SONALA-001 dosing
  PK for ALA and PpIX through 24 hours post SONALA-001 infusion: PK parameters for IV administered SONALA-001 and for the change in plasma concentration of the active metabolite PpIX will be estimated. Individual plasma concentrations will be listed by subject, summarized descriptively and graphically as warranted by drug dose and energy level. The following PK parameters will be calculated: AUC for plasma concentration vs. time from time 0 to the last measurable time point (AUC0-t), AUC for plasma concentration vs. time from time 0 to infinity (AUC0-∞), time to maximum drug concentration (Tmax), terminal elimination half-life (t½), clearance, and elimination rate constant.
To evaluate the mechanical performance of Exablate 4000 Type 2.0 device. | Day 1 to directly after each SDT treatment
  Mechanical performance of Exablate 4000 Type 2.0 device: Percentage of SDT treatments in which the Exablate 4000 Type-2 device works as planned and percentage of treatments in which procedure deviations were noted.

OTHER OUTCOMES:
To evaluate the safety and tolerability of SDT in the DMG subjects | Day 1 (SDT Study Treatment Day) to 12 months post-treatment
  Safety and tolerability as assessed by the frequency and severity of dose-limiting toxicities (DLTs), AEs, laboratory and ECG tests, vital signs, weight, physical and neurological exams
To evaluate the objective response rate (ORR) in the DMG subjects. | Day 1 to 12 months
  An estimate of RAPNO-ORR or mRANO-ORR, dependent on the age of the subject, will be derived as the percentage of subjects achieving a complete or partial response (CR, PR) relative to the total sample size in the full analysis set.
Progression-free survival (PFS) in the DMG subjects. | Day 1 to 12 months
  PFS is defined as the time from enrollment to the first progressive disease or all-cause mortality
Duration of response (DOR) in the DMG subjects. | Day 1 to 12 months
  The time-to-event under consideration in the analysis of DOR will be time from onset of (RAPNO) response to the time of first progression of disease.
Overall survival (OS) in the DMG subjects. | Day 1 to 24 months
  OS is defined as the time from enrollment to all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Corina Andresen, MD, Study Director — SonALAsense, Inc.
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Children's National / Children's Research Institute, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: No